CLINICAL TRIAL: NCT02529358
Title: Evaluation of a Transdiagnostic Text Message Based Maintenance Intervention After Inpatient Cognitive Behavioural Therapy
Brief Title: Text Message Based Maintenance Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Collaborators: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Dipl.-Psych. Sandra Schlicker, Dipl.-Psych., Friedrich-Alexander-Universität Erlangen-Nürnberg
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: SMS-MI
Record Dates: First submitted 2015-03-18; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Mental Disorders
Keywords: Maintenance intervention; Text messages; Emotion Regulation
MeSH Terms: conditions — Mental Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EG stand (Experimental): Standardized text messages
  Interventions: Behavioral: standardized text messages
- EG ind (Experimental): Personalized text messages
  Interventions: Behavioral: Personalized text messages
- Control (Other): Standardized text messages after 10 weeks
  Interventions: Behavioral: Standardized text messages after 10 weeks

INTERVENTIONS:
Behavioral: standardized text messages — Messages consist of relaxation techniques and mindfulness exercises as well as emotion regulation strategies
  Arms: EG stand
Behavioral: Personalized text messages — Patients write their own messages
  Arms: EG ind
Behavioral: Standardized text messages after 10 weeks — Messages consist of relaxation techniques and mindfulness exercises as well as emotion regulation strategies which are send to the patients 10 weeks after completing inpatient therapy
  Arms: Control

SUMMARY:
The study presents findings from a randomized clinical trial evaluating the effects of text messages encouraging short emotion regulation exercises on the course of psychopathological symptoms after inpatient treatment for depression. In this context, the study also compares the effectiveness of standardized versus personalized text messages.

DETAILED DESCRIPTION:
Introduction: The importance of aftercare and maintenance intervention to reduce psychopathology, prevent relapses and stabilize the effects of inpatient cognitive behavioral therapy is well proven. In order to attain a high reachability rate among the patients, simple, quick and low cost methods should be used. Modern communication technologies, such as mobile phones provide this opportunity. Therefore, the current study explores how modern communication technologies can be used as a support system in psychotherapy to realize a reduced psychopathology.

Methods: A total of 150 patients participated in a transdiagnostical 6-weeks text messaging maintenance intervention. The text messages were based on emotion regulation skills. The effectiveness of different variants of the text messages was studied in a randomized controlled trial, comparing the impact on the patient's psychopathological outcome to receiving personalized text messages versus standardized text messages.

ELIGIBILITY:
Inclusion Criteria:

* good knowledge of the german language
* owning a mobile phone

Exclusion Criteria:

* brain damage
* personality disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Depressive Symptom load | 6 weeks post treatment (after intervention)
  Measurement of depressive symptom severity with Beck Depression Inventory
Emotion Regulation Competence | 6 weeks post treatment (after intervention)
  Emotion Regulation Competence measured by SERSA

SECONDARY OUTCOMES:
Psychopathological symptomatology | 10 weeks Follow-Up
  Measurement of psychopathological symptomatology with self report questionnaires
Depressive Symptom load | 10 weeks Follow-Up
  Measurement of depressive symptom severity with Beck Depression Inventory
Emotion Regulation Competence | 10 weeks follow up
  Emotion Regulation Competence measured by SERSA

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Schlicker, Dipl.-Psych., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg; Matthias Berking, Prof. Dr., Study Chair — Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- Schön Klinik, Bad Arolsen, Hesse, Germany